CLINICAL TRIAL: NCT03634345
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, FIXED-SEQUENCE, PARALLEL-COHORT STUDY TO ESTIMATE THE EFFECT OF FLUVOXAMINE OR FLUCONAZOLE, ON THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF A SINGLE DOSE OF PF-04965842 IN HEALTHY SUBJECTS
Brief Title: Drug Drug Interaction Study Evaluating the Effect of Fluvoxamine or Fluconazole on PK and Safety of PF-04965842.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7451017; 2018-001943-29 (EudraCT Number)
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-04965842 (Experimental): investigational drug
  Interventions: Drug: Period 1 - Day 1: PF-04965842 administered; Drug: Period 2: Cohort 1: Fluvoxamine & PF-04965842; Drug: Period 2: Cohort 2: Fluconazole & PF-04965842

INTERVENTIONS:
Drug: Period 1 - Day 1: PF-04965842 administered — Period 1: Single administration of 100 mg PF 04965842.
  Other Names: Single administration of PF-04965842 in Period 1.
Drug: Period 2: Cohort 1: Fluvoxamine & PF-04965842 — Cohort 1: Period 2: Administration of fluvoxamine from Day 1 to Day 9 and PF-04965842 on Day 8.
  Other Names: 9-day administration of Fluvoxamine and single administration of PF-04965842 on day 8.
Drug: Period 2: Cohort 2: Fluconazole & PF-04965842 — Cohort 2: Period 2: Administration of fluconazole from Day 1 to Day 7 and PF-04965842 on Day 5.
  Other Names: 7-day administration of fluconazole and single administration of PF-04965842 on day 5.

SUMMARY:
A Phase 1, Open Label, Parallel-Cohort, Randomized, Fixed Sequence Study To Evaluate The Pharmacokinetic Drug Drug Interaction Between PF-04965842 and Fkuvoxamine (cohort 1) or Fluconazole (Cohort 2) in healthy subjects.

DETAILED DESCRIPTION:
A phase 1 study to evaluate the effect of fluvoxamine (a strong CYP2C19 and moderate CYP3A inhibitor) or fluconazole (a strong CYP2C19, moderate CYP2C9 and CYP3A inhibitor) on the pharmacokinetics, safety and tolerability of PF-04965842 in healthy subjects.

This study will be a Phase 1, open label, randomized, fixed-sequence, parallel-cohort study drug-drug interaction study. The study includes 2 periods:

In Period 1: all subjects will receive one single oral dose of 100 mg PF 04965842 tablet. (Treatment A). PK will be evaluated in the first 72 hours post adminstration of PF 04965842.

In Period 2:

* Cohort 1: subjects will receive fluvoxamine (immediate release tablet 50 mg) once daily for 9 consecutive days; on Day 8, subjects will receive a single oral dose of 100 mg PF 04965842 approximately 3 hours after fluvoxamine administration. (Treatment B). PK will be evaluated in the first 72 hours post administration of PF 04965842.
* Cohort 2: subjects will receive fluconazole capsule(s) once daily for 7 consecutive days (400 mg on Day 1 and 200 mg on Day 2-7 in Period 2); on Day 5, subjects will receive a single oral dose of 100 mg PF 04965842 approximately 1 hour after fluconazole administration. (Treatment C). PK will be evaluated in the first 72 hours post administration of PF 04965842.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Evidence or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination.
* History of hypersensitivity to or intolerance of fluvoxamine and/or fluconazole.
* Any condition possibly affecting drug absorption.
* A positive urine drug test.
* Screening supine systolic BP <90 mm Hg or 140 mm Hg following at least 5 minutes of supine rest OR Screening supine diastolic BP <50 mm Hg or 90 mm Hg following at least 5 minutes of supine rest.
* Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Plasma Cmax for PF 04965842 | First 72 hours post PF-04965842 administration in Period 1 and Period 2
  Maximum Observed Plasma Concentration (Cmax) for PF 04965842
AUCinf for PF-04965842 | First 72 hours post PF-04965842 administration in Period 1 and Period 2
  Area Under the Curve From Time Zero to Extrapolated Infinite Time for PF 04965842 (AUCinf)

SECONDARY OUTCOMES:
Number of subjects with Adverse events (AEs) | Screening up to 28 Days after the Last Dose of PF 04965842
  Number of subjects with Adverse events (AEs)
Number of subjects with laboratory tests findings of potential clinical importance | Screening up to 7-14 Days after the Last Dose of PF 04965842 in Period 2
  Number of subjects with laboratory tests findings of potential clinical importance
Number of Subjects with clinically significant abnormal Vital Signs | Screening up to 7-14 Days after the Last Dose of PF 04965842 in Period 2
  Number of Subjects with clinically significant abnormal Vital Signs
Number of Subjects with Electrocardiograms (ECGs) findings of potential clinical importance | Screening up to 7-14 Days after the Last Dose of PF 04965842 in Period 2
  Number of Subjects with Electrocardiograms (ECGs) findings of potential clinical importance

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang X, Dowty ME, Wouters A, Tatulych S, Connell CA, Le VH, Tripathy S, O'Gorman MT, Winton JA, Yin N, Valdez H, Malhotra BK. Assessment of the Effects of Inhibition or Induction of CYP2C19 and CYP2C9 Enzymes, or Inhibition of OAT3, on the Pharmacokinetics of Abrocitinib and Its Metabolites in Healthy Individuals. Eur J Drug Metab Pharmacokinet. 2022 May;47(3):419-429. doi: 10.1007/s13318-021-00745-6. Epub 2022 Feb 28. PMID 35226304
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451017&StudyName=A+Phase+1%2C+Open-label%2C+Randomized%2C+Fixed-sequence%2C+Parallel-cohort+Study+To+Estimate+The+Effect+Of+Fluvoxamine+Or+Fluconazole%2C+On+The+Pharmacokinetics%2C+Safety+And+Tolerability+Of+A+Single+Dose+Of+Pf-04965842+In+Healthy+Subjects